CLINICAL TRIAL: NCT01553552
Title: Comparison of Schistosomiasis Diagnostic Techniques and Study of Schistosoma Infection on Children's Immune Response to Childhood Vaccines, on Anaemia and on Nutritional Status
Brief Title: Schistosomiasis Effect on Response to Vaccines, Anaemia and Nutritional Status of Children of Northern Senegal
Acronym: SchistoVAN
Status: Completed | Type: Observational
Sponsor: Biomedical Research Center EPLS (Other)
Collaborators: Institut Pasteur de Lille (Other); University of Lille Nord de France (Other); Région Nord-Pas de Calais, France (Other); Centre d'Infection et d'Immunité de Lille (Other); Centre National de la Recherche Scientifique, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: EPLS11-MS
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Schistosomiasis; Anemia; Underweight; Stunting; Intestinal Parasites
Keywords: Schistosoma haematobium; schistosoma mansoni; Anemia; Underweight; stunting; Blastocystis
MeSH Terms: conditions — Schistosomiasis; Anemia; Thinness; Growth Disorders; Intestinal Diseases, Parasitic; Schistosomiasis haematobia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood Sera Urine Stool
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Infected by Schistosoma haematobium
- Not infected by Schistosoma haematobium

SUMMARY:
SchistoVAN aims to study the role of schistosomiasis infection in the modulation of the immune response of children to childhood vaccine antigens, as well as the impact of this infection on their nutritional status and their haemoglobinaemia.

DETAILED DESCRIPTION:
SchistoVAN aims to study the interactions between chronic parasite infections such as schistosomiasis and the immunological and nutritional status of children. In this scope, the investigators conducted a case-control study where one group of children is infected with schistosoma haematobium and the other is not infected with this parasite.

The investigators then stimulated whole blood of these children with various vaccine antigens to address their immune function and study the influence of schistosomiasis infectious state on their overall immune condition.

Aims of the study:

To evaluate the interaction between schistosomiasis and the nutritional status of children and their haemoglobinemia.

To evaluate the influence of schistosomiasis on children's specific immune response towards EPI vaccine antigens, the inflammatory status of children and nutritional serologic markers.

To compare schistosomiasis diagnostic tools (evaluation of circulating cathodic antigen (CCA) strip for diagnosis of urinary schistosomiasis in comparison with microscopy and urinary dipsticks)

To study prevalence of intestinal parasites such as Blastocystis hominis

ELIGIBILITY:
Inclusion Criteria:

* Members of AnoPalAnoVac cohort
* Age: between 6 and 10 years

Exclusion Criteria:

* body temperature > 38.5 ºC
* malaria episode

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Residents of 3 villages from the Senegal Valley River, belonging to the Podor District in Saint-Louis Region in Northern Senegal: Agniam Towguel, Fanaye Diery and Niandane. Subcohort of a previous study "AnoPalAnoVac" (ClinicalTrials.gov ID: NCT01545115)
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Hermann, PhD A.Pr., Study Chair — Biomedical Research Center EPLS; Lobna Gaayeb, VetMed, Study Director — Biomedical Research Center EPLS; Modou Seck, MD, Principal Investigator — Biomedical Research Center EPLS
Locations (1):
- Biomedical Research Center EPLS, Saint-Louis, SL, Senegal

REFERENCES:
- [Derived] Hermann E, Gaayeb L, Sow PS, Seck M, Sagna AB, Senghor S, Bandagny L, Brinkhuizen C, Delcroix-Genete D, Schacht AM, Riveau G. Sex-dependent interactions between leptin, wasting and humoral immunity in two ethnic communities of school-aged children differentially exposed to Schistosoma haematobium. Trans R Soc Trop Med Hyg. 2017 Oct 1;111(10):448-456. doi: 10.1093/trstmh/trx078. PMID 29351649
- See also: EPLS website — http://www.espoir-sante.org